CLINICAL TRIAL: NCT00665028
Title: Perioperative Ischemia Reduction Study (PROSE) Pilot
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: SpaceLab (Unknown); Research in Motion (Unknown); Globestar (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2007246-01H
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Myocardial Ischemia
Keywords: Anesthesia; Postoperative myocardial ischemia; ST monitoring
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Postoperative myocardial ischemia

SUMMARY:
After surgery, patients who have cardiogram changes consistent with a lack of oxygen to the heart muscles, also known as myocardial ischemia, have been found to have 9 times the chance of having an event such as a heart attack during the subsequent 30 days. It is not known if monitoring and treating ischemia will prevent events such as heart attacks. It is not known if such monitoring and treatment can be done on the regular surgical wards. In this pilot study, we hope to demonstrate that such a study is feasible, and the maintenance of blinding is possible. The primary outcomes are to show that such monitoring after surgery is possible in ≥ 95% of patients, to show that response and treatment to such ischemia in ≤ 1 hour is possible in ≥ 90% of patients, and that blinding between the standard and active treatment groups is possible for 50% ± 1 s.d.. With the pilot study data, if successful, we will be applying for peer-reviewed funding for a full study.

DETAILED DESCRIPTION:
Perioperative myocardial ischemia has been studied in the pre-, intra-, and postoperative periods. The intraoperative incidence is similar to the preoperative period but the postoperative incidence is doubled that of the preoperative period. These results have two implications: postoperative myocardial ischemia cannot be predicted by preoperative ambulatory ECG monitoring since only half of those are seen preoperatively; the postoperative period is when significant myocardial ischemia occurs.

The role of myocardial ischemia, especially prolonged ischemia, in perioperative myocardial infarction (PMI) has been recognized by a number of investigators. In the presence of postoperative myocardial ischemia, the relative risk of a postoperative cardiac event was 16 in one study and the odds ratio for an ischemic cardiac event was 9.2 in another. Using 12-lead continuous monitoring, one study found that all PMI were preceded by myocardial ischemia.

Ambulatory ECG in the postoperative period has been well reported in the past. Recently, Landesberg reported the sensitivity and specificity of lead placements to detect myocardial ischemia in the postoperative period. Lead combinations were compared with continuous 12-lead ECG in 185 consecutive patients. Combining two precordial leads, the sensitivity for detecting ischemia was 97.4% for V3 + V5; 92.1% for V4 + V5; and for infarction was 100% for V3 + V5 or V4 + V5.

We believe that the pathogenesis of PMI is multifactorial. Apart from the coronary anatomy and the vulnerable plaque, stress hormones and catecholamine surges in the perioperative period are well reported. Stress increases systolic BP, which is a major determinant of LV wall tension, and hence, myocardial oxygen demand. The oxygen cost of "pressure work" is greater than "volume work", with the area-under-the-curve for LV pressure closely correlating with myocardial oxygen demand. Hypercoagulable state has also been implicated in PMI.

With so many possible pathogenesis, it is our belief therefore that postoperative myocardial ischemia may be one of the final pathways just before postoperative ischemic cardiac complications. This is especially so when all PMI were preceded by myocardial ischemia in one study. With potentially multiple pathogenesis, it is unknown if postoperative myocardial ischemia is amenable to treatment. It is, however, our belief that postoperative myocardial ischemia can be aborted using existing treatment modalities. The implication is that the reduction of postoperative myocardial ischemia may reduce the incidence of postoperative ischemic cardiac complications, including PMI.

Current standard of care does not include telemetry or real-time ST monitoring on surgical patients. Traditional telemetry would impede low-risk patients in their postoperative recovery by limiting them to their beds. In the context of real-time monitoring for ST changes in low-risk patients, the cost of traditional telemetry with nursing may also be prohibitive. We propose a novel technological application, transmitting wireless ST segment monitoring and alarms to a Blackberry. This will alert the research team to verify via "full disclosure" on the ST monitor and respond directly. SpaceLab, GlobeStar, and Research in Motion (RIM) have developed the hardware and software respectively. We currently have written assurances and support from SpaceLab, GlobeStar, and RIM to conduct a pilot study for this novel application (see attached). We therefore propose a pilot study to determine the feasibility of wireless ST-segment monitoring and its treatment in post-surgical patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55 years
2. RCRI Class; 3 (i.e. 2 factors)
3. Elective non-cardiac surgical procedure
4. Expected to stay in hospital 2 days

Exclusion Criteria:

1. Atrial fibrillation
2. Left bundle branch block (LBBB)
3. Pacemaker dependency
4. Digoxin
5. CABG / PCI within 5 years
6. Low risk surgery (TURP, digit re-implantation, nerve repair, etc)
7. Expected ICU admission
8. CO2 retention
9. Refusal to transfusions
10. Adverse drug reaction to NSAIDS, beta-blockers, Ca-channel blockers, statins, nitrates
11. Prior enrolment in PROSE

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective non-cardiac surgical procedure
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Perioperative Ischemia Reduction Study Pilot (PROSE) & (PROSE 2) | 12 months
  Observational study on feasibility of remote ECG ST monitoring on a wireless system.
Feasibility of remote wireless ECG ST monitoring | 24 months
  To study the feasibility of real-time remote wireless ECG ST monitoring through wireless infrastructure of the hospital

CONTACTS AND LOCATIONS:
Overall Officials: H Yang, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada